CLINICAL TRIAL: NCT03582137
Title: A Randomized, Double Blind, Placebo-controlled Parallel Study of Tolerability and Efficacy of Cannabidiol (CBD) on Motor Symptoms in Parkinson's Disease
Brief Title: A Study of Tolerability and Efficacy of Cannabidiol on Motor Symptoms in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-2318
Record Dates: First submitted 2018-04-17; First posted 2018-07-10 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Motor symptoms; Tremor; tolerability; safety; cognition; anxiety; psychosis; mood; dyskinesia; sleep; cannabidiol; cannabis; efficacy; non-motor symptoms; quality of life; seborrhea
MeSH Terms: conditions — Parkinson Disease; Tremor; Anxiety Disorders; Psychotic Disorders; Dyskinesias; Marijuana Abuse; Dermatitis, Seborrheic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD Cannabis extract oral solution (Experimental): Cannabidiol (CBD) Cannabis extract oral solution
  Interventions: Drug: Cannabidiol
- placebo (Placebo Comparator): Placebo oral solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Subjects randomized to this arm will receive Cannabidiol Cannabis extract oral solution
  Other Names: CBD
  Arms: CBD Cannabis extract oral solution
Other: Placebo — Subjects randomized to this arm will receive Placebo
  Arms: placebo

SUMMARY:
The major purpose of this study is to assess the efficacy of CBD on motor symptoms of Parkinson's Disease (PD), and secondarily to study the safety and tolerability of CBD and other efficacy, particularly regarding tremor in PD. The study has been powered to detect a clinically significant reduction in Movement Disorder Society (MDS) Unified Parkinson's Disease Rating Scale (UPDRS) Part III motor scores. This is a 1:1 parallel, double-blind, randomized controlled trial (RCT) with 60 participants. The investigators will be recruiting up to 75 participants; the goal is to have 60 participants (30 in CBD group and 30 in placebo group) complete the study. The study drug is obtained from the National Institute on Drug Abuse (NIDA).

DETAILED DESCRIPTION:
Persons with PD have progressive disabling tremor, slowness, stiffness, balance impairment, cognitive deficits, psychiatric symptoms, autonomic dysfunction, fatigue and insomnia. Tremor may interfere with necessary daily and work functions. The disorder affects approximately seven million people globally. The total economic cost in the US is around 23 billion dollars. In addition to economic costs, PD reduces quality of life of those affected and their caregivers.

Cognitive impairment is a common feature and ranges from delayed recall in early stages to global dementia in up to 80% at end stage. PD with dementia has been associated with reduced quality of life, shortened survival, and increased caregiver distress. Community-based studies have estimated the point prevalence for dementia in PD to be 28% and 44%.

Depression, anxiety and psychosis are also common and are particularly disabling in PD, even at the earliest stages. These symptoms have important consequences for quality of life and daily functioning, are associated with increased carer burden and risk for nursing home admission. Anxiety affects up to 40% of patients with PD, and may predate motor symptoms by several years. The most common anxiety disorders in PD are panic attacks (often during off-periods), generalized anxiety disorder, and simple and social phobias. Psychotic symptoms vary in frequency according to the definition used. If mild forms are included, these affect up to 50% of patients. Visual hallucinations are the most common type. However, hallucinations occur in all sensory domains and delusions of various types are also relatively common. The impact of psychosis is substantial in that it is associated with dementia, depression, earlier mortality, greater caregiver strain, and nursing home placement. Thus, it is crucial to treat these symptoms in order to optimize the management of PD patients.

Generally, however, current therapies are inadequate. Medications have improved the prognosis of PD, but also have problematic adverse effects.

Since treatment of PD is often unsatisfactory and since cannabis has recently become legal and readily available in Colorado, persons with PD have been trying it. Patients have heard from the internet, support groups and other sources that marijuana is helpful. Most are doing so on their own, without the supervision or even knowledge of their neurologist. In a survey conducted in the spring of 2014 in University of Colorado Hospital Movement Disorders clinic about 5% of 207 PD patients, average age 69, reported using cannabis. In another study reported that 25% of PD patients had taken cannabis in the General University Hospital in Prague. In the investigators clinics, about 30% of the PD patients have asked doctors during their clinic visits over the past 6 months about cannabis. In an anonymous web-based survey, 72% PD patients reported current or past using medical cannabis, and 48% reducing prescription medication since beginning cannabis use.

PD mostly affects the elderly, and affected persons often have cognitive, psychiatric and motor problems, such as being prone to falling. Cannabis is well documented to cause psychosis, anxiety, slowness and incoordination. Studies have also shown that chronic users have structural and functional Central Nervous System (CNS) alterations. Thus cannabis is expected to be risky in persons with PD. Further, there are many components of cannabis, and the cannabis preparations being sold in Colorado vary widely in composition. There are no definitive data regarding the benefits and risks in of these various preparations in PD. Studies on safety and efficacy are greatly needed to protect this fragile Colorado population.

Human trials report that CBD decreases anxiety and causes sedation in healthy individuals, decreases psychotic symptoms in schizophrenia and PD, and improves motor and non-motor symptoms and alleviates levodopa-induced dyskinesia in PD. Given the current literature regarding CBD: possible neuroprotective effect, good tolerability, anxiolytic and antipsychotic effects and general lack of information in PD, including its effect on tremor, the investigators feel that it is important to study its use in PD further. The investigators hypothesized that it would reduce tremor, anxiety and psychosis, and would be well tolerated in PD.

The Specific Aims are:

Primary Specific Aim: To evaluate the efficacy of CBD on motor symptoms in PD, specifically on the motor section of the Movement Disorders Society Unified PD Rating Scale (MDS-UPDRS).

Secondary Specific Aim: To assess the safety and tolerability of CBD in PD, and to examine the effect of CBD on severity & duration of intractable tremor, night-time sleep, rigidity, emotional dyscontrol, anxiety and pain in PD.

Exploratory Analyses:

To study the efficacy of CBD on cognition, psychosis, sleep, daytime sleepiness, mood, fatigue, impulsivity, bladder function, other motor and non-motor PD signs, restless legs syndrome and Rapid Eye Movement (REM) sleep behavior disorder and quality of life. To explore the effect of CBD on plasma levels in PD.

The study is a randomized, placebo controlled, double-blind parallel design with two treatment arms, each of approximately 2-3 weeks duration. In the 2-3 week treatment phase participants will start study drug and titrate up to the maximum tolerated or targeted dose (2.5 mg/kg/day of CBD). Each participant will have a screening visit, baseline visit within 3 weeks, 1 liver function monitoring visits on 3rd to 5th day of 2.5 mg/kg/day, 2 dose assessment visit (1.25 mg/kg/day and 2.5 mg/kg/day), and a safety visit (6 visits total). Participants will be evaluated on the 3rd to 5th day at each dose level for monitoring liver function and adverse events, as well as changes in medical history and concomitant medications. Participants are called 3 days and 1 week after stopping the study drug to check for signs of withdrawal.

ELIGIBILITY:
Inclusion criteria:

* Male or female participants 40 - 85 years of age.
* Willing and able to give informed consent (including through use of a legally authorized representative (LAR), if necessary).
* Idiopathic PD, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* ON motor MDS UPDRS >20.
* Anti-parkinsonian medication is fixed for at least one month prior to the day the participant starts study drug treatment.
* If MoCA<22 participant must have a designated caregiver that agrees to ensure study protocols followed. This includes accompanying patient to study visits and being available for study phone calls.
* Must have a driver or available transportation (including provided Uber vouchers) to drive them to and from study visits and for other transportation needs during the treatment period.
* Has a significant other (someone who knows the participant well) that is appropriate for doing the NPI assessment, and agrees to do so
* Agrees to not take more than 1 gram per day of acetaminophen, due to a possible interaction with study drug that could increase risk of hepatotoxicity.

Exclusion criteria:

* Known or suspected allergy to cannabinoids or excipients used in the study drug formulation.
* Cannabis is detectable at the screening visit by blood testing or at the baseline visit by urine testing. If cannabis is detected at either the screening or baseline visit, then the participant is a screen fail and may return >14 days later for a repeat screening visit. If cannabis is again detected at either the screening or baseline visit, then the participant is excluded and not allowed to rescreen.
* History of drug or alcohol dependence; defined by prior inpatient stay(s) for this or that patient states s/he has a history of this.
* Use of dopamine blockers within 180 days and amphetamine, cocaine, and MAO-A inhibitors within 90 days of baseline.
* Currently taking tolcapone, valproic acid, felbamate, niacin (nicotinic acid) at ≥2000 mg/day or nicotinamide (nicotinic acid amide or nicotinamide) at ≥3000 mg/day, isoniazid and ketoconazole due to risk of liver injury and clobazam and ketoconazole because of risk of toxic interactions with the study drug. These medications need to be stopped 90 days before the baseline visit.
* Unstable medical condition.
* Any of the following laboratory test results at screening:

Hemoglobin < 10 g/dL WBC <3.0 x 109/L Neutrophils <1.5 x 109/L Lymphocytes < 0.5 x 109/L Platelets <100 x 109/L Hemoglobin A1C > 9%

* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal. Persons with stable liver disease of known etiology can be included, unless total bilirubin or prothrombin time/INR is abnormal.
* Is pregnant or lactating, or has a positive pregnancy test result pre-dose.
* If a sexually active female, is not surgically sterile or at least two years post-menopausal, or does not agree to utilize an effective method of contraception from screening through at least four weeks after the completion of study treatment, using one of the following: barrier methods (diaphragm or partner using condoms plus use of spermicidal jelly or foam, preferably double-barrier methods); oral or implanted hormonal contraceptive; intrauterine device (IUD); or vasectomized male partner.
* Planned elective surgery during study participation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Leehey, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available by request from qualified investigators who provide a valid research question, for 20 months after the trial is electronically published.
Supporting Information: Study Protocol, SAP
Time Frame: 20 months after the trial is electronically published.
Access Criteria: by request from qualified investigators who provide a valid research question; as approved by Principal Investigator

REFERENCES:
- [Derived] Weber I, Zagona-Prizio C, Sivesind TE, Adelman M, Szeto MD, Liu Y, Sillau SH, Bainbridge J, Klawitter J, Sempio C, Dunnick CA, Leehey MA, Dellavalle RP. Oral Cannabidiol for Seborrheic Dermatitis in Patients With Parkinson Disease: Randomized Clinical Trial. JMIR Dermatol. 2024 Mar 11;7:e49965. doi: 10.2196/49965. PMID 38466972

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between 9/5/2018 and 1/4/2022, 74 participants were screened, 61 randomized and 31 assigned to the CBD/THC drug and 30 to placebo. 13 participants were excluded: 8 participants not meeting inclusion criteria, and 5 declined to participate after screening.
Period: Overall Study
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Started | 31 | 30
Completed | 30 | 30
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (6.2) | 68.6 (7.6) | 69.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 18 | 23 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 28 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Disease duration [Mean (Standard Deviation); unit: years] | 7.0 (6.8) | 4.5 (3.9) | 5.8 (5.7)
Modified Hoehn & Yahr [Mean (Standard Deviation); unit: units on a scale] | 2.47 (0.69) | 2.30 (0.48) | 2.39 (0.61)
Baseline • Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part III [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS)- The MDS UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). Part III has instructions for the rater to give or demonstrate to the patient; it is completed by the rater. Scores ranges 0 -132. Higher values represent a worse outcome.
  units on a scale | 34.6 (9.1) | 30.9 (9.0) | 32.8 (9.3)
Baseline total Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS)- The MDS UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). Total score ranges 0-260. Higher values represent a worse outcome.
  units on a scale | 56.7 (17.9) | 48.8 (15.5) | 52.8 (17.4)
Levodopa-equivalent daily dosage [Mean (Standard Deviation); unit: mg/day] | 417.9 (440.3) | 427.5 (292.8) | 422.7 (370.7)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] | 26.9 (3.6) | 27.1 (2.2) | 27.0 (3.0)
Married [Count of Participants; unit: Participants] | 25 | 23 | 48
Retired [Count of Participants; unit: Participants] | 25 | 24 | 49
Education, >=college educated [Count of Participants; unit: Participants] | 23 | 27 | 50
Income >$75,000 [Count of Participants; unit: Participants] | 17 | 18 | 35
Body weight [Mean (Standard Deviation); unit: kg] | 79.0 (16.2) | 82.1 (12.4) | 80.5 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination) Scores
Description: Movement Disorders Society-Unified Parkinson's disease rating scale(MDS UPDRS) Part III assesses the motor signs of PD. There are 33 scores based on 18 items, several with right, left or other body distribution scores.Each question is anchored with five responses that are linked to commonly accepted clinical terms: 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe. The possible change may be the scores of the total 33 scores. Scores ranges 0 -132. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day of CBD, through 3 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
units on a scale | -4.5714 [-8.1126 to -1.0302] | -2.7665 [-4.9213 to -0.6118]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.3785, Mixed Models Analysis; Mean Difference (Net) = -1.8049, 95% CI 2-sided [-5.8839 to 2.2741]

2. Secondary Outcome: The Number of Participants Wtih Treatment-related Adverse Events
Description: Adverse events (AEs) are collected at each dose level. AEs collection include Serious Adverse Events (SAE), withdrawal symptoms and common AEs. SAE is an undesirable medical occurrence that results in death, or life-threatening, or inpatient hospitalization or prolongation of existing hospitalization or significant disability or incapacity or in a congenital anomaly/birth defect. Withdrawal and common AEs include headache, anxiety, nausea/vomiting, tremor, chills, decreased concentration, increased concentration, agitation, irritability, sleep disturbances, mood changes, somnolence, fatigue, anorexia, appetite changes, weight loss or gain, diarrhea, convulsion, abdominal pain, weakness, fever and other unexpected AEs. All of the these AEs will be recorded and counted.
Time Frame: Every 3-5 days at each dose level, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 26 | 25

3. Secondary Outcome: Change in Liver Function Monitoring --Liver Function Test
Description: Liver function tests will be performed and evaluated at each clinic visit from baseline through 3 weeks. The result is reported as the number of participants that had a clinically significant change in the values of the liver function test, including aspartate aminotransferase (AST), Alanine transaminase (ALT), Gamma-glutamyl transferase (GGT), Alkaline phosphatase (Alk Phos), Total Bilirubin (TB).
Time Frame: Baseline; at the end of 2.5 mg/kg/day; and every 3-5 days at each dose level, through 3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

4. Secondary Outcome: The Number of Participants Wtih Liver Function Impairment Related Adverse Events
Description: Liver function impairment will be evaluated and then related to adverse events and documented at each clinic visit. The change may be the frequency and severity of liver function impairment related AEs, including nausea/vomiting, diarrhea, abdominal pain, fatigue, weakness, chills, appetite changes, weight loss or gain, fever, etc.
Time Frame: Baseline; at the end of 2.5 mg/kg/day; and every 3-5 days at each dose level, through 3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants
  nausea | 6 | 3
  diarrhea | 2 | 4
  fatigue | 10 | 6
  abdominal pain | 1 | 3
  anorexia | 2 | 3
  weight loss | 1 | 2
  not applicable | 9 | 9

5. Secondary Outcome: Change in Blood Pressure (Systolic)
Description: Standing systolic blood pressure measurements will be assessed through 3 weeks. The change may be the value of systolic blood pressure.
Time Frame: Baseline; at the end of 2.5 mg/kg/day, through 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in mmHg
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in mmHg | -5.4145 [-11.4569 to 0.6279] | -0.9891 [-6.4615 to 4.4833]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.2712, Mixed Models Analysis; Mean Difference (Net) = -4.4254, 95% CI 2-sided [-12.4018 to 3.5510]

6. Secondary Outcome: Change in Vital Signs-heart Rate
Description: The change may be Heart rate (beat/minute) while standing.
Time Frame: Baseline; at the end of 2.5 mg/kg/day, through 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in beats per minute
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in beats per minute | 0.9459 [-3.1640 to 5.0559] | 0.6326 [-2.1185 to 3.3838]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.8974, Mixed Models Analysis; Mean Difference (Net) = 0.3133, 95% CI 2-sided [-4.5414 to 5.1680]

7. Secondary Outcome: Change in Vital Signs--weight
Description: The change may be weight in kilograms or lbs.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in kilograms
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in kilograms | 0.07389 [-0.2163 to 0.3641] | -0.07658 [-0.4177 to 0.2645]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.4643, Mixed Models Analysis; Mean Difference (Net) = 0.1505, 95% CI 2-sided [-0.2882 to 0.5892]

8. Secondary Outcome: Change in Vital Signs--temperature (Fahrenheit Degree)
Description: The change may be temperature in Fahrenheit degree
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in degrees Fahrenheit
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in degrees Fahrenheit | -0.3069 [-0.6335 to 0.01972] | -0.1882 [-0.5579 to 0.1816]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.6245, Mixed Models Analysis; Mean Difference (Net) = -0.1188, 95% CI 2-sided [-0.6019 to 0.3644]

9. Secondary Outcome: Change in Physical Exam
Description: The result is reported as the number of participants that had a clinically significant change in the physical exam findings, including allergic immunologic, cardiovascular, constitutional symptoms, ENT, endocrine, eyes, gastrointestinal, genitourinary, hematologic, integumentary, musculoskeletal, neurological, psychiatric, respiratory and other symptoms clinical significant findings.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

10. Secondary Outcome: Change in Neurological Exam
Description: The result is reported as the number of participants that had a clinically significant change in the general neurological exam clinical significant findings, including cranial nerves, motor strength, sensation, reflexes, gait, and other movements.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

11. Secondary Outcome: Change in Electrocardiograms
Description: The result is reported as the number of participants that had a clinically significant change in the EKG.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

12. Secondary Outcome: Change in Laboratory Values--hematology
Description: The result is reported as the number of participants that had a clinically significant change in the values of Hematology parameters, including RBC, WBC, HB, PLT, et al.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

13. Secondary Outcome: Change in Laboratory Values--chemistry
Description: The result is reported as the number of participants that had a clinically significant change in the values of the Chemistry profile, including BUN, CR, Electrolyte, glucose, liver function, etc.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

14. Secondary Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: Montreal Cognitive Assessment (MoCA) is a rapid screening instrument for mild cognitive dysfunction. The change may be the scores of MoCA, which is ranging from 0-30. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.8341 [-1.7743 to 0.1062] | -0.5000 [-1.3489 to 0.3489]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.5921, Mixed Models Analysis; Mean Difference (Net) = -0.3341, 95% CI 2-sided [-1.5749 to 0.9068]

15. Secondary Outcome: Change in Wechsler Test for Adult Reading
Description: The change may be the scores of Wechsler test for Adult Reading. Wechsler Test of Adult Reading (WTAR) - Word reading tests are an established method of establishing a premorbid estimate of verbal intellectual functioning, which will serve as an estimate of premorbid cognitive reserve. The WTAR comprises 50 words with irregular pronunciations that participants read aloud. The raw score can be transformed to an age-adjusted standard score, which is used to predict IQ (M = 100; SD = 15). Scores higher means better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: Out of the total study population, 25 participants took the cognitive test from CBD group, and 26 from placebo group.
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 25 | 26
change in units on a scale | 0.4421 [-1.6349 to 2.5192] | -1.4931 [-3.0859 to 0.09972]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution; Test type: Superiority; p = 0.1016, Mixed Models Analysis; Mean Difference (Net) = 1.9352, 95% CI 2-sided [-0.4372 to 4.3076]

16. Secondary Outcome: Change in Grooved Pegboard Test
Description: The change are the scores of Grooved Pegboard Test for the dominant affected hand. Manipulative dexterity, including finger speed, is assessed. Scoring is the time it took the participant to complete the task. Start the clock once the participant starts and stop it once the task has been completed. If after five minutes the participant has not completed the pegboard, stop the participant. The score the higher the worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: Out of the total study population, 15 participants performed the cognitive test from CBD group, and 14 from placebo group.
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 15 | 14
change in seconds | 5.3406 [-12.2701 to 22.9514] | -14.3454 [-27.0367 to -1.6540]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.0661, Mixed Models Analysis; Mean Difference (Net) = 19.6860, 95% CI 2-sided [-1.3733 to 40.7452]

17. Secondary Outcome: Change in Symbol Digit Modalities Test
Description: The change may be the scores of Intellectual functioning estimate, Symbol digit modalities test (SDMT). The SDMT is a measure of processing speed and working memory that has proven to be sensitive to cognitive impairment in MS that has both oral and written trials (only the oral trial will be administered given the anticipated difficulty patients will have with tremor). Participants are presented with a key at the top of a page pairing unique symbols with single digits. Participants are required to provide the correct digit with symbols that are presented on the rest of the page. The score is the number of correctly coded items from 0-110. The number of correct responses provided in 90 seconds on the oral trial is recorded. Scores range 0-110 items. The higher the score the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: Out of the total study population, 29 participants performed the cognitive test from CBD group, and 29 from placebo group.
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 29 | 29
change in units on a scale | 0.6143 [-2.0546 to 3.2832] | 3.8357 [1.1306 to 6.5408]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.0880, Mixed Models Analysis; Mean Difference (Net) = -3.2214, 95% CI 2-sided [-6.9381 to 0.4953]

18. Secondary Outcome: Change in Paced Auditory Serial Addition Test
Description: The change may be the scores of Intellectual functioning estimate, Paced auditory serial addition test. Paced Auditory Serial Addition Test (PASAT) - The PASAT is a more complex measure of processing speed and working memory in which a series of digits is presented to participants at varying intervals (i.e., 2 seconds, 3 seconds). Participants must add each digit to the immediately preceding digit for the duration of each trial. The number of correct responses for each trial is recorded. The score for the PASAT is the total number correct out of 60 possible answers. The higher, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: Out of the total study population, 27 participants performed the cognitive test from CBD group, and 25 from placebo group.
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 27 | 25
change in units on a scale | 6.9653 [-0.04668 to 13.9773] | 11.9489 [5.5760 to 18.3219]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.2827, Mixed Models Analysis; Mean Difference (Net) = -4.9836, 95% CI 2-sided [-14.2093 to 4.2421]

19. Secondary Outcome: Change in Controlled Oral Word Association Test
Description: The change may be the scores of Intellectual functioning estimate, Controlled oral word association test (COWAT). The COWAT is a measure of speeded verbal fluency and word retrieval in which participants are asked to say as many words as they can that begin with each of three letters for 60 seconds. The total number of words generated across all three trials is recorded. The higher, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 29 | 29
change in units on a scale | 3.1675 [1.0881 to 5.2470] | 2.5916 [-0.8430 to 6.0262]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.7703, Mixed Models Analysis; Mean Difference (Net) = 0.5760, 95% CI 2-sided [-3.3697 to 4.5216]

20. Secondary Outcome: Change in Hopkins Verbal Learning Test-total Learning
Description: The change may be the scores of Intellectual functioning estimate, Hopkins verbal learning test-revised. Hopkins Verbal Learning Test-Revised (HVLT-R) - The HVLT-R is a measure of verbal learning and memory in which participants are asked to learn a 12-item word list over three trials (total immediate learning). When scoring, the three leaning trials are combined to calculate a total recall score. Score ranges 0-36. The higher, the better. The outcoe measure is reporting the change from baseline in the total leaning score across all three trials.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: Out of the total study population, 26 participants performed the cognitive test from CBD group, and 25 from placebo group.
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 26 | 25
change in units on a scale | -2.03 (1.06) | -1.30 (1.15)
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.1874, Mixed Models Analysis; Mean Difference (Net) = -0.8834, 95% CI 2-sided [-2.2172 to 0.4504]

21. Secondary Outcome: Change From Baseline for the Delayed Recall Trials Score of HVLT-R
Description: Hopkins Verbal Learning Test-Revised (HVLT-R) Delayed recall trial. The participant is asked to recall as many words as they can 20-25 minutes after being presented the word list. The range is 0-12; the higher, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: as for outcome 20
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 26 | 25
change in units on a scale | -1.16 (0.60) | -0.28 (0.26)

22. Secondary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Delayed Recognition Trial
Description: The change may be the scores of Intellectual functioning estimate, Hopkins verbal learning test-revised. Hopkins Verbal Learning Test-Revised (HVLT-R) is a measure of verbal learning and memory in which participants are asked to learn a 12-item word list over three trials (total immediate learning). Delayed recognition trials is composed of 24 words, including the 12 target words and 12 false-positives, 6 semantically related, and 6 semantically unrelated. Retention % = percentage retained or delayed recall divided by better score on trial 2 or 3. Range 0-1. The higher, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: as for outcome 20
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale | 0.54 (0.48) | 0.55 (0.27)

23. Secondary Outcome: Change in Judgment of Line Orientation
Description: The change may be the scores of Intellectual functioning estimate, Judgment of line orientation. Judgment of Line Orientation (JOLO) - The JOLO is test of visuospatial functioning which measures a person's ability to match the angle and orientation of lines in space. Patients are asked to match two angled lines to a set of 11 lines that are arranged in a semicircle and separated 18 degrees from each other. Score ranges 0-30. The higher, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 26 | 25
change in units on a scale | 0.1367 [-1.0173 to 1.2907] | -1.1626 [-2.6697 to 0.3446]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.1646, Mixed Models Analysis; Mean Difference (Net) = 1.2993, 95% CI 2-sided [-0.5533 to 3.1519]

24. Secondary Outcome: Change in Semantic Verbal Fluency
Description: The change may be the scores of Semantic verbal fluency. Semantic Verbal Fluency - Semantic Verbal fluency is a measure of speeded verbal fluency and word retrieval in which participants are asked to say as many animal names/fruits and vegetables for 60 seconds. The total number of words generated across all three trials is recorded. The higher the score is, the better.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 29 | 29
change in units on a scale | 0.7153 [-0.7948 to 2.2253] | 2.4672 [0.8614 to 4.0729]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.1093, Mixed Models Analysis; Mean Difference (Net) = -1.7519, 95% CI 2-sided [-3.9082 to 0.4045]

25. Secondary Outcome: Change in Anxiety Short Form Response
Description: Comprised of 8 items which has five response options. Anxiety short form - is component of the Neurol-QOL (Quality of Life in Neurological Disorders) Measurement System, which is a collaborative effort of the National Institute of Neurological Disorders and Stroke and a number of partnering institutions. This measurement system was designed to be responsive to the needs of researchers in a variety of neurological disorders and to facilitate comparisons of data across clinical trials in different diseases. The short form is comprised of eight items that were selected from the respective item bank. Items have five response options (e.g., 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always). Respondents generally can answer five questions per minute. The change may be the total scores of the 8 items. Higher values represent a worse outcome. Scores range 8-40.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -2.1001 [-3.6111 to -0.5891] | -3.4533 [-4.8327 to -2.0740]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.1819, Mixed Models Analysis; Mean Difference (Net) = 1.3532, 95% CI 2-sided [-0.6511 to 3.3576]

26. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI)
Description: Valid and reliable scale to provide a means of assessing neuropsychiatric symptoms and psychopathology of patients. The change may be the scores of NPI. Neuropsychiatric Inventory (NPI) - is a valid and reliable scale. It was developed to provide a means of assessing neuropsychiatric symptoms and psychopathology of patients with Alzheimer's disease and other neurodegenerative disorders. It has proven to be sensitive to change and has been employed to capture treatment related behavioral. The NPI is administered to a caregiver/significant other who has detailed knowledge of the participant's behavior. Higher values represent a worse outcome. Score ranges 0-12.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in units on a scale | -0.3000 [-0.9611 to 0.3611] | -1.2667 [-2.7392 to 0.2058]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.2282, Mixed Models Analysis; Mean Difference (Net) = 0.9667, 95% CI 2-sided [-0.6287 to 2.5621]

27. Secondary Outcome: Change in Scales of Outcomes in Parkinson's Disease (SCOPA) Sleep-daytime Sleepiness
Description: Scales for Outcomes in Parkinson's disease (SCOPA)sleep - is a valid, reliable, short scale for assessing daytime sleepiness (DS) and nighttime sleep problems (NS) in patients with PD. The DS sub scale evaluates daytime sleepiness and includes six items with four response options, ranging from 0 (never) to 3 (often). The score ranges 0-18. The higher the worse. The other
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: 31 patients from CBD group and 30 from placebo group conducted the SCOPA DS scales.
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.5280 [-1.2572 to 0.2012] | -0.2667 [-1.0365 to 0.5031]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.6167, Mixed Models Analysis; Mean Difference (Net) = -0.2614, 95% CI 2-sided [-1.3002 to 0.7775]

28. Secondary Outcome: Change in Depression Short Form
Description: Comprised of 8 items which item has five response options. Depression short form - is a component of the Neurol-QOL (Quality of Life in Neurological Disorders) Measurement System, which is a collaborative effort of the National Institute of Neurological Disorders and Stroke and a number of partnering institutions. This measurement system was designed to be responsive to the needs of researchers in a variety of neurological disorders and to facilitate comparisons of data across clinical trials in different diseases. The short form is comprised of eight items that were selected from the respective item bank. Items have five response options (e.g., 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always). Respondents generally can answer five questions per minute.
  The change may be the scores of the total 8 items. Score ranges 0-40. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
change in units on a scale | -1.7300 [-3.9531 to 0.4931] | -2.0367 [-4.1183 to 0.04500]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.8378, Mixed Models Analysis; Mean Difference (Net) = 0.3067, 95% CI 2-sided [-2.6765 to 3.2899]

29. Secondary Outcome: Change in Emotional and Behavioral Dyscontrol Short Form
Description: Comprised of 8 items which item has 5 response options. Emotional and behavioral dyscontrol short form - is a component of the Neurol-QOL Measurement System, which is a collaborative effort of the National Institute of Neurological Disorders and Stroke and a number of partnering institutions. This measurement system was designed to be responsive to the needs of researchers in a variety of neurological disorders and to facilitate comparisons of data across clinical trials in different diseases. The short form is comprised of eight items that were selected from the respective item bank. Items have five response options (e.g., 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always). Respondents generally can answer five questions per minute.
  The change may be the total scores of the 8 items. Score ranges 0-40. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -3.9870 [-6.3219 to -1.6522] | -4.2733 [-6.8021 to -1.7445]

30. Secondary Outcome: Change in Stanford Sleepiness Scale
Description: Is a quick and easy way to assess how the participant is feeling. The change may be the scores of the scale 3 hours after dosing compared to pre-dosing.
  Stanford Sleepiness Scale (SSS): The Stanford Sleepiness Scale is a quick and easy way to assess how alert the participant is feeling. SSS is validated and probably the most widely used instrument for the assessment of participant's sleepiness.
  Score ranges 0-7. Higher values represent a worse outcome.
Time Frame: Pre- and 3 hours post- dose at baseline visit
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | 0.2903 [-0.1380 to 0.7187] | -0.03333 [-0.3298 to 0.2631]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.2103, Mixed Models Analysis; Mean Difference (Net) = 0.3237, 95% CI 2-sided [-0.1880 to 0.8353]

31. Secondary Outcome: Change in Pain Intensity 3a Short Form
Description: Assess how much a person hurts. The change may be the score of the short form. Pain Intensity 3a short form - components of the Patient Reported Outcome Measurement Information System (PROMIS), which was developed by the NIH to provide a standardized metric for measuring physical, mental, and social health across chronic diseases. PROMIS instruments were developed using item response theory and have been tested in more than 20,000 individuals drawn from the general US population. The Pain Intensity instrument assesses how much a person hurts. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Each question has five response options ranging in value from one to five.
  Score ranges 0-15. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -3.1209 [-4.9451 to -1.2968] | -2.6169 [-4.8111 to -0.4226]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.7197, Mixed Models Analysis; Mean Difference (Net) = -0.5040, 95% CI 2-sided [-3.3015 to 2.2934]

32. Secondary Outcome: Change in Pain Interference 4a Short Form
Description: Self-reported consequences of pain on relevant aspects of one's life. The change may be the scores of the short form.
  The Pain Interference instrument measures the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Each question has five response options ranging in value from one to five.
  Score ranges 0-20. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.1543 [-2.1498 to 1.8412] | -2.7701 [-4.8473 to -0.6929]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.0686, Mixed Models Analysis; Mean Difference (Net) = 2.6158, 95% CI 2-sided [-0.2058 to 5.4373]

33. Secondary Outcome: Change in Fatigue Severity Scale
Description: Self-report 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity. The change may be the total scores of the 9 items, ranging from 9-63. Higher values represent worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | 1.4224 [-2.2727 to 5.1175] | -1.3667 [-4.3254 to 1.5920]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.2339, Mixed Models Analysis; Mean Difference (Net) = 2.7891, 95% CI 2-sided [-1.8523 to 7.4304]

34. Secondary Outcome: Change in Movement Disorder Society Unified Parkinson Disease Rating Scale
Description: Movement Disorder Society Unified Parkinson Disease Rating Scale. There are four parts, non-motor experiences of daily living, motor experiences of daily living, motor examination, and motor complications. The change may be the total scores of the four parts. Total score ranges 0-260. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -6.2798 [-11.5293 to -1.0303] | -7.2333 [-10.5756 to -3.8911]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.7557, Mixed Models Analysis; Mean Difference (Net) = 0.9536, 95% CI 2-sided [-5.1655 to 7.0727]

35. Secondary Outcome: Change in Unified Dyskinesia Rating Scale
Description: To evaluate involuntary movements often associated with treated PD. The change may be the total scores of the scale, including historical sub-score (0-60) and objective sub-score (0-44). The total score is historical sub score plus objective sub score, ranged from 0- 104. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: In CBD group, 31 patients at baseline and 29 patients at 2.5 mg/kg/day were testes. In Placebo group, 30 at baseline and 28 at 2.5 mg/kg/day were tested.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 1.4704 [-1.4078 to 4.3487] | -1.4270 [-3.2753 to 0.4214]

36. Secondary Outcome: Change in the Timed UP&GO (TUG)
Description: The Timed Up & Go (TUG) test is a physical performance measure in which the ability to rise up from a seated chair position, walk 3m, turn, walk back, and sit down is timed. This measure is useful in an outpatient setting, because it requires only a few minutes, is easy to administer, and requires little equipment. Importantly, the TUG test is highly correlated with functional mobility, gait speed, and falls in older adults. The change may be the time duration (seconds) of performing the task. The higher, the worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
seconds | -0.5409 [-1.3780 to 0.2962] | -0.5922 [-1.0932 to -0.09113]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9150, Mixed Models Analysis; Mean Difference (Net) = 0.05126, 95% CI 2-sided [-0.9086 to 1.0111]

37. Secondary Outcome: Change in IRLS
Description: International restless legs syndrome (IRLS) study group rating scale for restless legs syndrome. The change may be the scores of the IRLS, ranged from 0-40. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -1.2366 [-3.3440 to 0.8709] | -0.5667 [-2.2772 to 1.1439]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.6164, Mixed Models Analysis; Mean Difference (Net) = -0.6699, 95% CI 2-sided [-3.3316 to 1.9918]

38. Secondary Outcome: Change in Rapid Eye Movement Sleep Behavior Disorder Screening Questionnaire (RBDSQ)
Description: REM sleep behavior disorder screening questionnaire (RBDSQ). The change may be the total scores of RBDSQ.
  REM sleep behavior disorder screening questionnaire (RBDSQ) - is a 10-item, patient self-rating instrument assessing the participant's sleep behavior with short questions that have to be answered by either "yes" or "no". Items 1 to 4 address the frequency and content of dreams and their relationship to nocturnal movements and behavior. Item 5 asks about self-injuries and injuries of the bed partner. Item 6 consists of four sub items assessing nocturnal motor behavior more specifically, e.g., questions about nocturnal vocalization, sudden limb movements, complex movements, or bedding items that fell down. Items 7 and 8 deal with nocturnal awakenings. Item 9 focuses on disturbed sleep in general and item 10 on the presence of any neurological disorder. The maximum total score of the RBDSQ is 13 points.
  Score ranges 0-13 points. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.4692 [-1.0392 to 0.1009] | -0.3333 [-1.0095 to 0.3429]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.7550, Mixed Models Analysis; Mean Difference (Net) = -0.1358, 95% CI 2-sided [-1.0028 to 0.7312]

39. Secondary Outcome: Change in Overactive Bladder Symptom Score
Description: A validated self-administered questionnaire consisting of 7 questions on a 5-point Likert scale. The change may be the scores of the scale, ranged from 0-35. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.09605 [-1.0385 to 0.8464] | 0 [-1.2663 to 1.2663]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9016, Mixed Models Analysis; Mean Difference (Net) = -0.09605, 95% CI 2-sided [-1.6449 to 1.4528]

40. Secondary Outcome: Change in Parkinson's Disease Questionnaire (PDQ-39)
Description: A reliable valid responsive acceptable and feasible tool for assessment of quality of life in PD, including 39 multiple-choice items covering 8 dimensions: mobility (#1-10), activities of daily living (#11-16), emotional well-being (#17-22), stigma (#23-26), social support (#27-29), cognition (#30-33), communication (#34-36), and bodily discomfort (#37-39). 5-point ordinal scoring system: 0=never, 1= occasionally, 2=sometimes, 3=often, 4=always. The change may be the total scores of PDQ-39, ranged from 0-156. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -4.8005 [-10.0155 to 0.4145] | -4.4788 [-8.6298 to -0.3278]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9219, Mixed Models Analysis; Mean Difference (Net) = -0.3217, 95% CI 2-sided [-6.8584 to 6.2151]

41. Secondary Outcome: Change in EuroQol-5 Dimension-5 Level
Description: Consists of 2 pages-the EuroQol-5 Dimension-5 level (EQ-5D-5L) descriptive system and the EuroQol (EQ) Visual analogue scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The VAS records the patient's self-rated health on a vertical visual analogue-scale, where the endpoints are labelled the best health you can imagine and the worst health you can imagine. The change may be the scales of EQ-5D. Score ranges 11111-55555. The higher, the worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | 0.05364 [0.009875 to 0.09741] | 0.02467 [-0.01451 to 0.06384]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.3178, Mixed Models Analysis; Mean Difference (Net) = 0.02897, 95% CI 2-sided [-0.02857 to 0.08651]

42. Secondary Outcome: Difference in Proportion of Participants That Discontinue the Study Due to Study Drug Intolerance
Description: Difference in Proportion of participants that discontinue the study due to study drug intolerance. The change may be the number of patients dropped out.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 1 | 0

43. Secondary Outcome: Change in Total Scores on Items 3.17 and 3.18 in MDS-UPDRS
Description: Rest tremor amplitude and constancy of rest tremor scores in MDS UPDRS. The change may be the sum scores of 3.17 and 3.18. Score ranged from 0-24. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -1.1570 [-2.0377 to -0.2763] | -0.1000 [-0.7625 to 0.5625]

44. Secondary Outcome: Change in Item 2.10 in MDS UPDRS
Description: Patient's tremor experience. The change may be the scores of item 2.10. Score ranged from 0-4. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.2280 [-0.4929 to 0.0368] | -0.100 [-0.3008 to 0.1008]

45. Secondary Outcome: Change in Item 3.15 and 3.16 in MDS UPDRS
Description: Postural tremor of the hands and kinetic tremor of the hand. The change may be the sum scores of item 3.15 and 3.16. Score ranged from 0-16. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.4291 [-0.9259 to 0.0677] | -0.6667 [-1.1317 to -0.2016]

46. Secondary Outcome: Change in Rigidity Sub Scores in MDS UPDRS
Description: Rigidity sub scores in MDS UPDRS. The change may be the sub scores of rigidity related item in MDS UPDRS (item 3.3). Score ranged from 0-20. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.3742 [-1.6096 to 0.8612] | -0.6030 [-1.5951 to 0.3891]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.7693, Mixed Models Analysis; Mean Difference (Net) = 0.2288, 95% CI 2-sided [-1.3250 to 1.7825]

47. Secondary Outcome: Change in Bradykinesia Sub Scores in MDS UPDRS
Description: Bradykinesia sub scores in MDS UPDRS. The change may be the sub scores of bradykinesia related items in MDS UPDRS, including items 3.4-3.8, and 3.14. The scores ranged from 0-44. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -1.6787 [-3.6134 to 0.2560] | -0.8666 [-2.6253 to 0.8921]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.5285, Mixed Models Analysis; Mean Difference (Net) = -0.8121, 95% CI 2-sided [-3.3743 to 1.7501]

48. Secondary Outcome: Change in Axial Sub Scores in MDS UPDRS
Description: Axial sub scores in MDS UPDRS. The change may be the sub scores of axial related items in MDS UPDRS, including items 3.9, 3.13, 3.10, 3.11, and 3.12. The sub scores ranged from 0-20. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.2919 [-0.8076 to 0.2237] | -0.2667 [-0.8275 to 0.2941]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9463, Mixed Models Analysis; Mean Difference (Net) = -0.02525, 95% CI 2-sided [-0.7717 to 0.7212]

49. Secondary Outcome: Change in Bulbar Sub Scores in MDS UPDRS
Description: Bulbar sub scores in MDS UPDRS (item 3.1 and 3.2). The change may be the sub scores of bulbar related items in MDS UPDRS, ranged from 0-8. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.3376 [-0.8015 to 0.1263] | -0.03333 [-0.6754 to 0.6088]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.4362, Mixed Models Analysis; Mean Difference (Net) = -0.3042, 95% CI 2-sided [-1.0817 to 0.4732]

50. Secondary Outcome: Change in Insomnia Severity Index
Description: Insomnia Severity Index (ISI): ISI is a verified seven-item self-report questionnaire assessing the nature, severity, and impact of insomnia. A five-point Likert scale is used to rate each item (e.g., 0=no problem; 4=very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
  A total score ranging from 0 to 28. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -1.6982 [-2.8162 to -0.5803] | -1.6333 [-2.7246 to -0.5421]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9327, Mixed Models Analysis; Mean Difference (Net) = -0.06489, 95% CI 2-sided [-1.5957 to 1.4659]

51. Secondary Outcome: Change in Pittsburgh Sleep Quality Index
Description: To measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. The change may be the total scores, ranged from 0 to 42. The higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.8226 [-1.7676 to 0.1225] | -1.5000 [-2.1722 to -0.8278]

52. Secondary Outcome: Change in Dermatology Quality of Life Index
Description: Dermatology quality of life index. The change may be the scores of the questionnaire. The scoring of each question is as follows: very much=3, a lot =2, a little=1, not at all=0, not relevant =0. Question 7, prevented work or studying =3. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.1763 [-0.7571 to 0.4044] | 0.1000 [-0.3343 to 0.5343]

53. Secondary Outcome: Change in the Number of Participants With Presence of Seborrheic Dermatitis From Baseline to Final Visit.
Description: Dermatology photography evaluation. The change in number of participants with a presence of seborrheic dermatitis from baseline to final visit. Dermatology photography: take a picture of the central face, as this is the most common area of seborrhea, and send it, with appropriate privacy safeguards, to dermatologists, Dr. Robert Dellavalle, MD., and Dr. Andrea Steel.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Number; unit: participants
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 29 | 29
participants | 2 | 3
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.4401, Mixed Models Analysis; Mean Difference (Net) = -0.2763, 95% CI 2-sided [-0.9880 to 0.4354]

54. Secondary Outcome: Change in Non-motor Symptoms Scale for Parkinson's Disease (NMSS)
Description: Validated 30-item scale for the assessment of NMS in PD. Each symptom scored with respect to severity (0=none, 1=mild, 2=moderate, 3=severe), frequency (1=rarely, 2=often, 3=frequent, 4=very frequent). Each NMSS item score is calculated by multiplying the severity and frequency score. The final score is the sum of the total 30-item scores. The change may be the total scores of NMSS, ranged from 0 to 360. The higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -5.8652 [-11.6281 to -0.1023] | -5.0333 [-8.9647 to -1.1020]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.8085, Mixed Models Analysis; Mean Difference (Net) = -0.8319, 95% CI 2-sided [-7.6835 to 6.0197]

55. Secondary Outcome: Change in Scales of Outcomes in Parkinson's Disease (SCOPA) - Daytime Sleep (DS) Problems.
Description: Scales for Outcomes in Parkinson's disease (SCOPA) sleep DS subscale is a valid, reliable, short scale for assessing daytime sleep problems (DS) in patients with PD. The sub scale includes six items with four response options, ranging from 0 (never) to 3 (often). The score ranges 0-18. The higher the worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: 31 patients from CBD group and 30 from placebo group conducted the SCOPA DS scales.
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -0.5280 (0.3575) | -0.2667 (0.3769)

56. Secondary Outcome: Change in Scales of Outcomes in Parkinson's Disease (SCOPA) - Nighttime Sleep (NS) Problems.
Description: Scales for Outcomes in Parkinson's disease (SCOPA) sleep NS subscale - is a valid, reliable, short scale for assessing nighttime sleep problems (NS) in patients with PD. The NS sub scale includes five items with four response options, ranging from 0 (never) to 3 (often). The score ranges 0-15. The higher the worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: 31 patients from CBD group and 30 from placebo group conducted the SCOPA NS scales.
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 31 | 30
change in units on a scale | -1.2066 (0.5075) | -1.2333 (0.4074)
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.9674, Mixed Models Analysis; Mean Difference (Net) = 0.02673, 95% CI 2-sided [-1.2757 to 1.3292]

57. Secondary Outcome: Change in Modified Dysfunctional Beliefs and Attitudes About Sleep Questionnaire (DBAS-16)
Description: Modified Dysfunctional Beliefs and Attitudes about Sleep Questionnaire (DBAS-16): A validated self-reported questionnaire designed to identify and assess various sleep/insomnia-related cognitions (e.g., beliefs, attitudes, expectations, appraisals, attributions). range is 0-160; the higher numbers are worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | -2.70 (3.40) | -4.57 (3.30)

58. Secondary Outcome: Change in Wake After Sleep Onset
Description: WASO, the total number of minutes that a person is awake after having initially fallen asleep; higher numbers are worse.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in minutes
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 21 | 25
change in minutes | -48.89 [-80.25 to -17.53] | -1.97 [-53.29 to 49.35]
Statistical Analysis 1: Comparison: CBD Cannabis Extract Oral Solution vs Placebo; Test type: Superiority; p = 0.1128, Mixed Models Analysis; Mean Difference (Net) = -46.92, 95% CI 2-sided [-105.51 to 11.68]

59. Secondary Outcome: Difference of Plasma Interleukin 6 Level Between PD and Healthy Control Population
Description: Interleukin 6 is an inflammatory cytokine, and is measured in the blood. Whole bold was collected into tubes containing anticoagulant; tubes were inverted gently 3-4 times. Blood was allowed to clot at room temperature for 30 to 45 min, centrifuged at 1,000 x g for 15 min at 4°C and serum was transferred to a clean polypropylene tube. To completely remove platelets and precipitates, the tubes were centrifuge again at 10,000 x g for 10 min at 4°C. Processed samples were stored at -80°F, and cytokine levels measured using the Bio-Plex ProTM Human Cytokine Assay.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Population: PD participants who took either cannabidiol cannabis extract oral solution or placebo.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- CBD Cannabis Extract Oral Solution; Placebo: Plasma cytokine levels were obtained from a subset of persons with PD excluding those with pre-existing abnormal inflammatory function: persons on chemotherapeutic, anti-inflammatory (including NSAIDS) and antihistaminic medications in the prior week, and that had active cancer, inflammatory or atopic conditions, or was being treated for any of these. This included any infection, for example the common cold or a urinary tract infection in the past week. In addition, persons with kidney failure or renal dialysis, uncontrolled heart disease, chronic respiratory disease requiring oxygen or medication, uncontrolled diabetes, active or treated seizures, and hyperthyroidism were excluded.
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 17 | 19
ng/mL | 2.99 [0.61 to 14.66] | 1.59 [0.33 to 7.66]

60. Secondary Outcome: Change in Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale (QUIP-RS) - Total Scores
Description: To measure severity of symptoms and support a diagnosis of impulse control disorders and related disorders in PD. The result is the difference of the change of the total scores of QUIP-RS (excessive hobbies-punding and dopamine dysregulation syndrome) between groups. The total QUIP-RS scores is 0-112. Higher values represent a worse outcome.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 29 | 30
score on a scale | -0.24 [-12 to 4] | 0.43 [0 to 8.00]

61. Secondary Outcome: Change in The Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a suicidal ideation rating scale. The change may be the answers to the questions of C-SSRS. There are five questions and have binary responses (yes/no). Assign a score of 1 if answer yes and score of 0 if no . Higher values represent a worse outcome.The mximum score is 5.
Time Frame: From baseline to the end of 2.5 mg/kg/day, assessed up to 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Adverse events are collected at all contacts with participants: primarily and formally at scheduled study visits (using a form) and phone calls (using a script), but also informally at any unscheduled contacts.
Arm/Group | CBD Cannabis Extract Oral Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/30
Other Adverse Events (participants affected / at risk) | 26/31 | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBD Cannabis Extract Oral Solution (N=31) | Placebo (N=30)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBD Cannabis Extract Oral Solution (N=31) | Placebo (N=30)
dizziness (Nervous system disorders) | 18 (18) | 6 (6)
feeling of relaxation (Nervous system disorders) | 13 (13) | 7 (7)
fatigue (Nervous system disorders) | 10 (10) | 6 (6)
decreased concentration (Nervous system disorders) | 10 (10) | 4 (4)
headache (Nervous system disorders) | 9 (9) | 10 (10)
somnolence (Nervous system disorders) | 8 (8) | 8 (8)
feeling abnormal (Nervous system disorders) | 8 (8) | 2 (2)
feeling drunk (Nervous system disorders) | 7 (7) | 2 (2)
nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
confusion (Nervous system disorders) | 5 (5) | 1 (1)
thinking abnormal (Nervous system disorders) | 5 (5) | 0 (0)
disorientation (Nervous system disorders) | 4 (4) | 0 (0)
dry mouth (General disorders) | 4 (4) | 1 (1)
fall (General disorders) | 4 (4) | 3 (3)
increased concentration (Nervous system disorders) | 4 (4) | 1 (1)
weakness (General disorders) | 4 (4) | 1 (1)
agitation (Nervous system disorders) | 3 (3) | 1 (1)
elevated mood (Nervous system disorders) | 3 (3) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4)
anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
anxiety (Nervous system disorders) | 2 (2) | 3 (3)
insomnia (Nervous system disorders) | 2 (2) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
sleep disturbance (Nervous system disorders) | 1 (1) | 2 (2)
weight loss (General disorders) | 1 (1) | 2 (2)
cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
depression (Nervous system disorders) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
chills (General disorders) | 2 (2) | 0 (0)
increased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
irritability (Psychiatric disorders) | 2 (2) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03582137/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT03582137/ICF_001.pdf